CLINICAL TRIAL: NCT04830384
Title: Evaluation Into the Efficacy of Low Level Laser/Light and Music as a Combined Therapy Device for Smoking Cessation Treatment
Brief Title: Evaluation of LLLT/Music for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Freedom Laser, Inc. (Industry)
Collaborators: NST Consultants, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLA1020
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Nicotine Dependence, Cigarettes
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Not all participants in this study will receive the actual, fully functioning device. One-quarter of the subjects will receive a fully functioning device with laser and music; one-quarter will receive laser only; one-quarter will receive music only; one quarter will receive a placebo or inactive device.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Fully Active (Experimental): LLLT & Music Therapy
  Interventions: Device: Fully Active
- LLLT Only (Active Comparator): LLLT Therapy
  Interventions: Device: LLLT Only
- Music Only (Placebo Comparator): Music Therapy
  Interventions: Device: Music Only
- Placebo (Sham Comparator): No Therapy
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Fully Active — 7 subjects will be dispensed active treatment devices with light and music fully functional
  Arms: Fully Active
Device: LLLT Only — 7 subjects will be dispensed active treatment devices with only light functional
  Arms: LLLT Only
Device: Music Only — 7 subjects will be dispensed placebo comparator devices with only music functional
  Arms: Music Only
Device: Placebo — 7 subjects will be dispensed placebo or sham devices with no light or music functional
  Arms: Placebo

SUMMARY:
The purpose of this research is to study the preliminary effectiveness of a light therapy and music device for at-home use to aid the seasoned cigarette smoker in his/her attempt to stop smoking. This device, called the FQS system, is a type of cold, or non-heat producing laser and tranquil music system that will emit light and music onto the ear surface, through commonly found music earphones, available in most electronic stores. The theory behind this treatment technique is that the light and music will stimulate the part of the brain responsible for producing chemicals that satisfy the desire for nicotine. If this is correct, then the user will replace the need for nicotine with the pleasant treatment experience of light and music therapy.

DETAILED DESCRIPTION:
This study aims to define the safety and physiologic effects that occur when low level light and music, configured in a wearable binaural head set are employed by seasoned smokers of cigarettes, with the end result of reducing the desire to smoke. This device use does not require any complementary or adjunctive drug use. A review of unregulated products that are marketed for smoking cessation, have as common mechanism of action, the administration and withdrawal of nicotine in a controlled dosing format. The proposed study device does not consider the use of the culprit drug, the best pathway to achieve rapid and long-lasting cessation results. The theoretical principle at work is the competition for absorption by nicotinic cholinergic receptors located in the brain by nicotine or by the LLLT and music therapy. If this competition for absorption by two competing elements (cigarettes and the proposed device) can result in the device "winning the race", then the neurotransmitters will respond to the LLLT and music stimulus instead of the serum nicotine and yield a reduced desire to consume nicotine. As with any new technology, it is essential to learn the variance between true efficacy and the placebo level of efficacy. This study seeks to define that variance.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects who have been smoking cigarettes for at least 5 years without any intervention therapy within the past 12 months.
* Apparent good health.
* Must admit to possessing the desire to stop smoking.
* Willing to use the proposed device at home, every day, for 15 minutes, for up to 6 weeks.
* Willing to participate in weekly monitoring program conducted through brief phone survey not to exceed 5 minutes per week.

Exclusion Criteria:

* Previous involvement in other smoking cessation studies.
* Use of any product, drug or device, designated as smoking cessation or reduction aid during the trial period or within the preceding last 12 months.
* Active and chronic consumption of any psychotropic or illicit drugs
* Evidence of any current viral, fungal or bacterial infection.
* Diagnosed mental disorders or habits that indicate self-destructive behavior, such as nail biting, morbid obesity, compulsive gambling or alcoholism.
* History of having been arrested for a criminal act or repeated non-criminal violations related to motor vehicle use.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Nicotine Consumption | 6 weeks
  Number of Cigarettes Smoked Daily

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Blanche, Study Director — NST Consultants, Inc.; Adam Bodian, MD, Principal Investigator — The Bodian Dermatology Group; Rebecca Settar, RN, Study Director — NST Consultants, Inc.
Locations (1):
- NST Consultants, Inc., Mendham, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No